CLINICAL TRIAL: NCT03557372
Title: Mathematical Model-Adapted Radiation Fractionation Schedule for Patients With Recurrent Glioblastoma (MARS-Glio)
Brief Title: Mathematical Model-Adapted Radiation In Glioblastoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Shyam Tanguturi, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-105
Record Dates: First submitted 2018-05-23; First posted 2018-06-15 (Actual); Results first posted 2021-06-11 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Recurrent Glioblastoma
Keywords: Recurrent glioblastoma; Radiation Therapy
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Mathematical Model-Adapted Radiation (Experimental): Mathematical Model-Adapted Radiation Fractionation Schedule
  Interventions: Radiation: Mathematical Model-Adapted Radiation Fractionation Schedule

INTERVENTIONS:
Radiation: Mathematical Model-Adapted Radiation Fractionation Schedule — * Re-irradiation with 35 Gy delivered over 2 weeks, based upon reference dosing of 35 Gy in 10 Fractions over 2 weeks
  * Radiation therapy is delivered on Monday-Friday during standard clinic hours in our department. Each treatment may take 20-40 minutes.
  * Treatment will be once daily for the first 7 days of treatment and then three-times daily for the last three days of treatment.

SUMMARY:
This research study is studying a new schedule of radiation therapy for recurrent glioblastoma as a possible treatment for this diagnosis. This radiation schedule is based on a new model for radiation resistance in glioblastoma.

The name of the radiation schedule involved in this study is:

- Re-irradiation for glioblastoma using a novel Mathematical Model-Adapted Radiation Fractionation Schedule

DETAILED DESCRIPTION:
This research study is a Feasibility Study, which means that this is the first time that investigators are examining this new radiation schedule for recurrent glioblastoma.

* The FDA (the U.S. Food and Drug Administration) has approved radiation therapy as a treatment option for your disease.
* This is the first time that this particular radiation schedule will be tested in humans. There many other studies which have tested different radiation schedules in glioblastoma.

In this research study, investigators are adapting a standard two-week schedule of radiation commonly used for recurrent glioblastoma using a mathematical model. This study uses the same total dose of radiation as standard treatments but breaks up the dose into different amounts daily to maximize tumor kill. investigators have used a new mathematical model to create this schedule of radiation. This model was created to better represent how glioblastoma cells can escape the damaging effects of radiation. Based on the results of several laboratory studies, it is possible that this model may result in improved outcomes compared to standard radiation schedules.

The primary question of this study is to see whether participants can complete this new radiation schedule at the scheduled times. In addition, investigators will follow participants to ensure that this treatment is safe. If this treatment proves feasible, investigators hope to compare this treatment directly with standard radiation schedules for newly diagnosed and recurrent glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have recurrent glioblastoma (WHO Grade IV), as defined on brain imaging with CT or MRI, after prior receipt of definitive therapy including neurosurgical biopsy or resection and radiation therapy with or without systemic therapy.
* Participants must be deemed appropriate candidates for re-irradiation
* Histopathologic confirmation of disease as part of routine clinical care is required either at the time of initial diagnosis and/or at the time of recurrent disease. There is no requirement for central pathologic review.
* Age ≥ 18 years at the time of enrollment
* Karnofsky Performance Status (KPS) of at least 70
* Exclusion Criteria
* Participants who have received more than one prior course of radiotherapy to the local site of progressive disease
* Participants who have received prior radiotherapy to the local site of progressive disease within < 3 months of the anticipated start of re-irradiation
* Participants with recurrent tumor extensively abutting or involving the optic structures or brainstem, as assessed by the treating radiation oncologist
* Participants without a definable tumor cavity on MRI or CT obtained at study enrollment
* Participants receiving concurrent cytotoxic chemotherapy (i.e. temozolomide, CCNU, vincristine, procarbazine) or concurrent immunotherapy (i.e. pembrolizumab, nivolumab); however, participants may receive sequential chemotherapy before or after radiation without limitation. Participants may receive concurrent corticosteroid and/or anti-angiogenic therapy (i.e. bevacizumab) if clinically indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2022-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Tanguturi, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Result] Dean JA, Tanguturi SK, Cagney D, Shin KY, Youssef G, Aizer A, Rahman R, Hammoudeh L, Reardon D, Lee E, Dietrich J, Tamura K, Aoyagi M, Wickersham L, Wen PY, Catalano P, Haas-Kogan D, Alexander BM, Michor F. Phase I study of a novel glioblastoma radiation therapy schedule exploiting cell-state plasticity. Neuro Oncol. 2023 Jun 2;25(6):1100-1112. doi: 10.1093/neuonc/noac253. PMID 36402744

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There are no details to report.
Groups:
- Mathematical Model-Adapted Radiation: Mathematical Model-Adapted Radiation Fractionation Schedule
  Mathematical Model-Adapted Radiation Fractionation Schedule: - Re-irradiation with 35 Gy delivered over 2 weeks, based upon reference dosing of 35 Gy in 10 Fractions over 2 weeks
  * Radiation therapy is delivered on Monday-Friday during standard clinic hours in our department. Each treatment may take 20-40 minutes.
  * Treatment will be once daily for the first 7 days of treatment and then three-times daily for the last three days of treatment.
Period: Overall Study
Arm/Group | Mathematical Model-Adapted Radiation
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants were counted for the primary endpoint of the study based on if they were able to complete the protocol specified course of radiation treatment or not.
Arm/Group | Mathematical Model-Adapted Radiation
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants to Complete Model Adapted Radiations Fractionation Scheduled
Description: Successful completion of radiotherapy is defined as receipt of all scheduled fractions of daily radiotherapy within 24 hours of once daily fractions and within 1 hour of three-times daily fractions.
Time Frame: 10 Days
Population: All 14 participants were analyzed for the primary endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Mathematical Model-Adapted Radiation
Number analyzed (Participants) | 14
Participants | 14

2. Secondary Outcome: Number of Participants With Radiation Necrosis
Description: Radiation necrosis (RN) was defined by clinical assessment including imaging features of an expansile, centrally hypointense lesion with increasing surrounding vasogenic edema and typically without features of high grade recurrence (restricted diffusion, elevated cerebral blood volume). Symptomatic RN included patients with radiographic RN requiring intervention such as corticosteroid therapy for neurologic symptoms, headaches, or signs of elevated intracranial pressure.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mathematical Model-Adapted Radiation
Number analyzed (Participants) | 14
Participants | 0

3. Secondary Outcome: Number of Participants With Seizures
Description: Count of number of patients developing new/worsening seizures within 6 months of receiving protocol radiation therapy
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mathematical Model-Adapted Radiation
Number analyzed (Participants) | 14
Participants | 1

4. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
Time Frame: range of follow-up from date of registration was 1.2 - 38.6 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Mathematical Model-Adapted Radiation
Number analyzed (Participants) | 14
Months | 7.3 [4.7 to 10.7]

5. Secondary Outcome: Grade 3-5 Treatment-related Toxicity Rate
Description: All grade 3-5 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv5 as reported on case report forms were counted. Rate is the proportion of treated participants experiencing at least one treatment-related grade 3-5 AE of any type during the time of observation.
Time Frame: 6 Months
Measure: Number; unit: proportion of treated participants
Arm/Group | Mathematical Model-Adapted Radiation
Number analyzed (Participants) | 14
proportion of treated participants | 0.29

6. Secondary Outcome: Median Progression-Free Survival (PFS)
Description: Progression-free survival based on the Kaplan-Meier method is defined as the duration between randomization and documented disease progression (PD) (defined protocol section 12.7) or death, or is censored at time of last disease assessment.
Time Frame: Disease evaluated on visit 4,5,6 and every 2-4 months in long-term. The range of follow-up from date of registration was 1.2 - 38.6 months and the median was 7.3 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Mathematical Model-Adapted Radiation
Number analyzed (Participants) | 14
Months | 4.3 [2.4 to 5.2]

7. Secondary Outcome: Median Local Recurrence-free Survival
Description: Local recurrence-free survival based on the Kaplan-Meier method is defined as the duration between randomization and documented Local recurrence or death, or is censored at time of last disease assessment.
Time Frame: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Mathematical Model-Adapted Radiation
Number analyzed (Participants) | 14
Months | 6.2 [5.2 to 30]

8. Secondary Outcome: Number of Participants Undergoing Salvage Craniotomy
Description: Count of patients undergoing salvage craniotomy for resection or decompression of progressively enlarging tumor within 6 months of receipt of protocol radiation therapy.
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Mathematical Model-Adapted Radiation
Number analyzed (Participants) | 14
Participants | 0

9. Secondary Outcome: Number of Participants Receiving Additional Systemic Treatments After Reirradiation
Description: Count of patients undergoing systemic therapies for presumed recurrence or progression of disease within 6 months after receipt of protocol radiation therapy
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Mathematical Model-Adapted Radiation
Number analyzed (Participants) | 14
Participants | 3

ADVERSE EVENTS:
Time Frame: Time-frame for observation of adverse events was up to 6 months of clinical follow up, and for all cause-mortality, up to 38.6 months.
Description: Serious adverse events (AEs) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv5. All remaining events regardless of treatment attribution were classified as Other AEs. Maximum grade toxicity by type for a patient over time was calculated. No further data is available to specify classification of other beyond the general term.
Arm/Group | Mathematical Model-Adapted Radiation
All-Cause Mortality (participants affected / at risk) | 13/14
Serious Adverse Events (participants affected / at risk) | 8/14
Other Adverse Events (participants affected / at risk) | 8/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mathematical Model-Adapted Radiation (N=14)
Death NOS (General disorders) | 8 (8)
Seizure (Nervous system disorders) | 1 (1)
Edema cerebral (Nervous system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mathematical Model-Adapted Radiation (N=14)
Nausea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Edema cerebral (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Quality of life assessment using MDASI-BT was incomplete due to patient preference and incomplete adherence. As such, assessment by this endpoint was not possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/72/NCT03557372/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT03557372/ICF_001.pdf